CLINICAL TRIAL: NCT05293158
Title: Impact of Hepatitis B Immunoglobulins in Patients With Chronic Hepatitis B on Hepatocellular Carcinoma
Brief Title: Impact of Hepatitis B Immunoglobulins in Patients With Chronic Hepatitis B on Hepatocellular Carcinoma - a Proof of Concept Study
Acronym: HBIG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBIG
Record Dates: First submitted 2022-03-14; First posted 2022-03-24 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma; HBV
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBIG treatment (Experimental)
  Interventions: Drug: Hepatect CP 50 I.E./ml infusion solution

INTERVENTIONS:
Drug: Hepatect CP 50 I.E./ml infusion solution — Application of i.v. (intravenously) HBIGs for ≥6-weeks:
  Day (D) 0-7: 10.000 IU D14 until end-of-treatment: 10.000 IU once per week HBIGs will be given until LT/liver resection.

SUMMARY:
In the current literature, infection with the hepatitis B virus (HBV) is described as one of the main risk factors for the development of hepatocellular carcinoma (HCC).

According to the current study situation, the Hepatitis B surface antigen (HBsAg) is considered as an important marker, since low levels and sero-clearance of HBsAg are both correlated with a lower risk of HCC development / recurrence.Currently there is no treatment option available that efficiently targets HBsAg. Besides neutralizing infectious HBV virions, Hepatitis B immunoglobulins (HBIG) can directly bind and neutralize extracellular HBsAg/SVPs, and even intracellular HBsAg targeting is reported. In addition, HBIGs can initiate effector-cell attack (via antibody-dependent cellular cytotoxicity, ADCC) towards infected hepatocytes.

The potential benefit of HBIGs in the HCC context is further underlined by recent evidence for the ability of HBIGs to reduce the viability, proliferation, and self-renewal of tumor-initiating cells (TICs) - isolated from HBV-HCC patients - accompanied by downregulation of stemness markers, e.g., OCT-4.According to the current study situation, the use of HBIGs significantly reduces the risk of HBV reinfection after transplantation and improves the results of liver transplantation in patients with chronic HBV infection. The potential benefit of treating HBV-HCC patients on the LTx (liver transplantation) waiting list with hepatitis B immunoglobulin is the possible stop or inhibition of tumor progression while waiting for an LTx. So far there is no clinical evidence of this.

Mechanistically, hepatitis B immunoglobulin could occur through neutralization of circulating HBsAg, which is an important driver of an immunosuppressive environment in HBV patients, and possibly through direct effects against HBV HCC tumor cells (through antibody-dependent cellular cytotoxicity, ADCC). Therefore, the idea behind preoperative HBIG administration before liver transplantation is to reduce the rate of patients in whom a transplantation would no longer have been possible due to tumor progression. Thus, due to tumor progression in HBV-positive HCC-patients there is a monthly drop-out from the waiting list of about 4%.

The basic idea behind the treatment of HBV-HCC patients before tumor resection with hepatitis B immunoglobulin is to potentially stop or positively influence tumor progression through the effects mentioned above, in the time between diagnosis and resection.

Zhou et al. (2015) have shown a connection between HBsAg levels and HCC relapses after resection, although the exact role of HBsAg is still unclear. In no case will the treatment postpone the time of tumor resection, as only patients are considered who, for clinical reasons, can expect a certain time until resection. The present proof of concept study aims to quantify HBsAg reduction due to preoperative administration of HBIGs in HBV-positive HCC-patients and serve as a template for future multicentre clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years and ≤ 80 of age
* HBsAg-positive HCC-patients scheduled for resection in ≥6 weeks or HBsAg-positive HCC- patients listed for LT
* Ability of subjects to understand character and individual consequences of the clinical trial
* Written informed consent must be available before enrolment in the trial

Exclusion Criteria:

* Clinically significant illness (other than HBV) or any other major medical disorder that, in the opinion of the investigator, may interfere with subject treatment
* No eligibility for resection / LT
* Concurrent any other malignancy
* Co-infection with hepatitis C virus (defined as HCV RNA positive, HCV RNA-negative/anti-HCV-positive patients can be included) and/or human immunodeficiency virus (HIV)
* Clinical hepatic decompensation
* Allergy to HBIG
* Pregnant, lactating patients

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
HBsAg change from baseline to week 6 | ≥6-weeks
  Quantification of the magnitude of the effect of ≥6-week; unit: IU/ml treatment with Hepatitis B immunoglobulins in patients with chronic hepatitis B and HCC, determined by the HBsAg reduction after week 6
  Evaluation of the safety and tolerability of Hepatitis B immunoglobulins administered for ≥6-weeks in patients with chronic hepatitis B and HCC

SECONDARY OUTCOMES:
Change of HBsAg at different time points during treatment | baseline and weekly during the treatment period and during the follow-up at 2 weeks, 4 weeks, 6 weeks, and 8 weeks after treatment stop.
  unit: IU/ml
Change of HCC response to treatment | Tumor material will be measured at baseline and at end of treatment (on average ≥6-weeks)
  Tumor size (cm) will be investigated via MR Primovist (RECIST) or alternatively via CT (RECIST).
Change of Biochemical response (B cells) | baseline and weekly during the treatment period and during the follow-up at 2 weeks, 4 weeks, 6 weeks, and 8 weeks after treatment stop.
  Immune responses during HBIG treatment (analysis of B cells); unit 10^9/l
Change of Biochemical response (NK cells) | baseline and weekly during the treatment period and during the follow-up at 2 weeks, 4 weeks, 6 weeks, and 8 weeks after treatment stop.
  Immune responses during HBIG treatment (analysis of NK cells); unit 10^9/l
Change of Biochemical response (T cells) | baseline and weekly during the treatment period and during the follow-up at 2 weeks, 4 weeks, 6 weeks, and 8 weeks after treatment stop.
  Immune responses during HBIG treatment (analysis of T cells); unit 10^9/l
Change of Cellular response (CD3) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (CD3); unit:10^9/L
Change of Cellular response (CD4) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (CD4); unit:10^9/L
Change of Cellular response (CD8) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (CD8); unit:10^9/L
Change of Cellular response (CD25) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (CD25); unit:10^9/L
Change of Cellular response (CD34) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (CD34); unit:10^9/L
Change of Cellular response (CD133) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (CD133); unit:10^9/L
Change of Cellular response (CD19) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (CD19); unit:10^9/L
Change of Cellular response (CD56) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (CD56); unit:10^9/L
Change of Cellular response (CD49f) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (CD49f); unit:10^9/L
Change of Cellular response (FoxP3) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (FoxP3) unit: µg/ml
Change of Cellular response (Ki67) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (Ki67) unit: %
Change of Cellular response (HLA-DR) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (HLA-DR) unit: %
Change of Cellular response (IFN gamma) | Tumor material will be collected at baseline and end-of-treatment (on average ≥6-weeks) via liver biopsies and will be analysed by immune histochemistry
  Tumor material will be collected via liver biopsies and will be analysed by immune histochemistry (IFN gamma) unit: IU/ml

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salpini R, Surdo M, Warner N, Cortese MF, Colledge D, Soppe S, Bellocchi MC, Armenia D, Carioti L, Continenza F, Di Carlo D, Saccomandi P, Mirabelli C, Pollicita M, Longo R, Romano S, Cappiello G, Spano A, Trimoulet P, Fleury H, Vecchiet J, Iapadre N, Barlattani A, Bertoli A, Mari T, Pasquazzi C, Missale G, Sarrecchia C, Orecchini E, Michienzi A, Andreoni M, Francioso S, Angelico M, Verheyen J, Ceccherini-Silberstein F, Locarnini S, Perno CF, Svicher V. Novel HBsAg mutations correlate with hepatocellular carcinoma, hamper HBsAg secretion and promote cell proliferation in vitro. Oncotarget. 2017 Feb 28;8(9):15704-15715. doi: 10.18632/oncotarget.14944. PMID 28152517
- [Background] Liu S, Koh SS, Lee CG. Hepatitis B Virus X Protein and Hepatocarcinogenesis. Int J Mol Sci. 2016 Jun 14;17(6):940. doi: 10.3390/ijms17060940. PMID 27314335
- [Background] Lee EC, Kim SH, Lee SD, Park H, Lee SA, Park SJ. High-dose hepatitis B immunoglobulin therapy in hepatocellular carcinoma with hepatitis B virus-DNA/hepatitis B e antigen-positive patients after living donor liver transplantation. World J Gastroenterol. 2016 Apr 14;22(14):3803-12. doi: 10.3748/wjg.v22.i14.3803. PMID 27076765
- [Background] Yang Y, Sun JW, Zhao LG, Bray F, Xiang YB. Quantitative evaluation of hepatitis B virus mutations and hepatocellular carcinoma risk: a meta-analysis of prospective studies. Chin J Cancer Res. 2015 Oct;27(5):497-508. doi: 10.3978/j.issn.1000-9604.2015.10.05. PMID 26543337
- [Background] Liu WR, Tian MX, Jin L, Yang LX, Ding ZB, Shen YH, Peng YF, Zhou J, Qiu SJ, Dai Z, Fan J, Shi YH. High levels of hepatitis B surface antigen are associated with poorer survival and early recurrence of hepatocellular carcinoma in patients with low hepatitis B viral loads. Ann Surg Oncol. 2015 Mar;22(3):843-50. doi: 10.1245/s10434-014-4043-5. Epub 2014 Oct 1. PMID 25269529
- [Background] Saab S, Yeganeh M, Nguyen K, Durazo F, Han S, Yersiz H, Farmer DG, Goldstein LI, Tong MJ, Busuttil RW. Recurrence of hepatocellular carcinoma and hepatitis B reinfection in hepatitis B surface antigen-positive patients after liver transplantation. Liver Transpl. 2009 Nov;15(11):1525-34. doi: 10.1002/lt.21882. PMID 19877207
- [Background] Lin S, Hoffmann K, Schemmer P. Treatment of hepatocellular carcinoma: a systematic review. Liver Cancer. 2012 Nov;1(3-4):144-58. doi: 10.1159/000343828. PMID 24159579
- [Background] Honer Zu Siederdissen C, Cornberg M. The role of HBsAg levels in the current management of chronic HBV infection. Ann Gastroenterol. 2014;27(2):105-112. PMID 24733569
- [Background] Tseng TC, Liu CJ, Yang HC, Su TH, Wang CC, Chen CL, Kuo SF, Liu CH, Chen PJ, Chen DS, Kao JH. High levels of hepatitis B surface antigen increase risk of hepatocellular carcinoma in patients with low HBV load. Gastroenterology. 2012 May;142(5):1140-1149.e3; quiz e13-4. doi: 10.1053/j.gastro.2012.02.007. Epub 2012 Feb 11. PMID 22333950
- [Background] Zahner D, Glimm H, Matono T, Churin Y, Herebian D, Mayatepek E, Kohler K, Gattenlohner S, Stinn A, Tschuschner A, Roderfeld M, Roeb E. Hepatitis B virus surface proteins accelerate cholestatic injury and tumor progression in Abcb4-knockout mice. Oncotarget. 2017 Feb 2;8(32):52560-52570. doi: 10.18632/oncotarget.15003. eCollection 2017 Aug 8. PMID 28881751
- [Background] Pollicino T, Cacciola I, Saffioti F, Raimondo G. Hepatitis B virus PreS/S gene variants: pathobiology and clinical implications. J Hepatol. 2014 Aug;61(2):408-17. doi: 10.1016/j.jhep.2014.04.041. Epub 2014 May 5. PMID 24801416
- [Background] Liu H, Xu J, Zhou L, Yun X, Chen L, Wang S, Sun L, Wen Y, Gu J. Hepatitis B virus large surface antigen promotes liver carcinogenesis by activating the Src/PI3K/Akt pathway. Cancer Res. 2011 Dec 15;71(24):7547-57. doi: 10.1158/0008-5472.CAN-11-2260. Epub 2011 Oct 12. PMID 21994334
- [Background] Churin Y, Roderfeld M, Roeb E. Hepatitis B virus large surface protein: function and fame. Hepatobiliary Surg Nutr. 2015 Feb;4(1):1-10. doi: 10.3978/j.issn.2304-3881.2014.12.08. PMID 25713800
- [Background] Li YW, Yang FC, Lu HQ, Zhang JS. Hepatocellular carcinoma and hepatitis B surface protein. World J Gastroenterol. 2016 Feb 14;22(6):1943-52. doi: 10.3748/wjg.v22.i6.1943. PMID 26877602
- [Background] Zhang X, Gao L, Liang X, Guo M, Wang R, Pan Y, Liu P, Zhang F, Guo C, Zhu F, Qu C, Ma C. HBV preS2 transactivates FOXP3 expression in malignant hepatocytes. Liver Int. 2015 Mar;35(3):1087-94. doi: 10.1111/liv.12642. Epub 2014 Aug 8. PMID 25047684
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] de Man RA, Metselaar HJ, Heijtink RA, Schalm SW. Long-term application of human polyclonal hepatitis-B immunoglobulin to prevent hepatic allograft infection. A review of the literature and presentation of five cases. Neth J Med. 1993 Aug;43(1-2):74-82. PMID 8232699
- [Background] Schilling R, Ijaz S, Davidoff M, Lee JY, Locarnini S, Williams R, Naoumov NV. Endocytosis of hepatitis B immune globulin into hepatocytes inhibits the secretion of hepatitis B virus surface antigen and virions. J Virol. 2003 Aug;77(16):8882-92. doi: 10.1128/jvi.77.16.8882-8892.2003. PMID 12885906
- [Background] Shouval D, Samuel D. Hepatitis B immune globulin to prevent hepatitis B virus graft reinfection following liver transplantation: a concise review. Hepatology. 2000 Dec;32(6):1189-95. doi: 10.1053/jhep.2000.19789. No abstract available. PMID 11093723
- [Background] Chang TS, Chen CL, Wu YC, Liu JJ, Kuo YC, Lee KF, Lin SY, Lin SE, Tung SY, Kuo LM, Tsai YH, Huang YH. Inflammation Promotes Expression of Stemness-Related Properties in HBV-Related Hepatocellular Carcinoma. PLoS One. 2016 Feb 26;11(2):e0149897. doi: 10.1371/journal.pone.0149897. eCollection 2016. PMID 26919045
- [Background] Beckebaum S, Herzer K, Bauhofer A, Gelson W, De Simone P, de Man R, Engelmann C, Mullhaupt B, Vionnet J, Salizzoni M, Volpes R, Ercolani G, De Carlis L, Angeli P, Burra P, Dufour JF, Rossi M, Cillo U, Neumann U, Fischer L, Niemann G, Toti L, Tisone G. Recurrence of Hepatitis B Infection in Liver Transplant Patients Receiving Long-Term Hepatitis B Immunoglobulin Prophylaxis. Ann Transplant. 2018 Nov 13;23:789-801. doi: 10.12659/AOT.910176. PMID 30420590
- [Background] Dindoost P, Jazayeri SM, Alavian SM. Hepatitis B immune globulin in liver transplantation prophylaxis: an update. Hepat Mon. 2012 Mar;12(3):168-76. doi: 10.5812/hepatmon.832. Epub 2012 Mar 28. PMID 22550524
- [Background] Cornberg M, Wong VW, Locarnini S, Brunetto M, Janssen HLA, Chan HL. The role of quantitative hepatitis B surface antigen revisited. J Hepatol. 2017 Feb;66(2):398-411. doi: 10.1016/j.jhep.2016.08.009. Epub 2016 Aug 27. PMID 27575311
- [Background] Thi Vo T, Poovorawan K, Charoen P, Soonthornworasiri N, Nontprasert A, Kittitrakul C, Phumratanaprapin W, Tangkijvanich P. Association between Hepatitis B Surface Antigen Levels and the Risk of Hepatocellular Carcinoma in Patients with Chronic Hepatitis B Infection: Systematic Review and Meta-Analysis. Asian Pac J Cancer Prev. 2019 Aug 1;20(8):2239-2246. doi: 10.31557/APJCP.2019.20.8.2239. PMID 31450890